CLINICAL TRIAL: NCT03054142
Title: China Collaborative Study on Epidemiology of Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: XinLing Liang (Other)
Responsible Party: Sponsor-Investigator, XinLing Liang, Director of Division of Nephrology and Blood Purification Center of Guangdong General Hospital, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Other Study IDs: CCS-AKI RF2011-2016
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AKI
  Interventions: Other: no intervention
- non-AKI
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Acute kidney injury (AKI) is a common clinical syndrome, especially patients in the hospital. AKI has become a huge medical burden in China. Little information is available about this disease burden in our country. The investigators aimed to evaluate the burden of AKI and to analyze the related risk factors.

DETAILED DESCRIPTION:
The investigators launch a nationwide of all patients, who were admitted to hospital from 2011-2016. Patients were diagnosed on the basis of changes in serum creatinine by the laboratory information system. The investigators assessed rates of AKI according to the criteria of 2012 Kidney Disease Improving Global Outcomes (KDIGO).

ELIGIBILITY:
Inclusion Criteria:

* The patients diagnosed on the basis of changes in serum creatinine according to the criteria of 2012 Kidney Disease Improving Global Outcomes(KDIGO)

Exclusion Criteria:

* Serum creatinine record less than two times during hospitalization
* Patients being diagnosed with End-stage kidney disease (chronic kidney disease stage 5)
* Nephrectomy
* Kidney transplantation
* Peak serum creatinine of less than 53µ mol/L
* Serum creatinine decrease after amputation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All inpatients (if outpatient identification is achieved, outpatient and inpatient patients can be judged to be the same individual, the outpatient electronic data is extracted at the same time)
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2017-01; Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AKI | Jan. 2011 to Oct. 2016

SECONDARY OUTCOMES:
Recognition rate of AKI | Jan. 2011 to Oct. 2016
  Using machine learning and deep learning methods to establish AKI prediction model and risk models
Proportion of nephrology referral | Jan. 2011 to Oct. 2016
In-hospital mortality | Jan. 2011 to Oct. 2016
Longer ICU stay | Jan. 2011 to Oct. 2016
Higher medical cost | Jan. 2011 to Oct. 2016

CONTACTS AND LOCATIONS:
Overall Officials: Liang Xinling, M.D.,Ph.D, Principal Investigator — Nephrology Dept,Guangdong General Hospital
Locations (1):
- Nephrology Dept,Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu L, Wu Y, Chen Y, Li R, Wang Z, Li Z, Liu G, Yu L, Shi W, Liang X; China collaborative study on AKI (CCS-AKI). Is acute kidney injury age-dependent in older adults: an observational study in two centers from North China. BMC Geriatr. 2021 Jan 6;21(1):7. doi: 10.1186/s12877-020-01906-z. PMID 33407184